CLINICAL TRIAL: NCT04716309
Title: Unstable Distal Radius Fractures AO-type A2, A3 and C1 With Dorsal Dislocation in Patients Aged 18-64 Years. Open Reduction and Volar Locking Plate Versus Closed Reduction and Percutaenous Pinning. A Randomized Controlled Trial.
Brief Title: Unstable Distal Radius Fractures With Dorsal Dislocation in Patients Aged 18-64 Years. Volar Locking Plate (VLP) vs Closed Reduction and Percutaenous Pinning (CRPP).
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sophies Minde Ortopedi (Industry)
Responsible Party: Principal Investigator, Børge Olsen, MD Børge Olsen, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 85724
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Distal Radius Fractures; Wrist Fracture; Colles' Fracture
MeSH Terms: conditions — Wrist Fractures; Colles' Fracture | interventions — Open Fracture Reduction; Bone Wires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLP (Active Comparator): Open reduction and volar locking plate
  Interventions: Procedure: Open reduction and volar locking plate and closed reduction and K-wires.
- CRPP (Active Comparator): Closed reduction and percutaenous K-wires/pins
  Interventions: Procedure: Open reduction and volar locking plate and closed reduction and K-wires.

INTERVENTIONS:
Procedure: Open reduction and volar locking plate and closed reduction and K-wires. — DVR Anatomic Plate, K-wires

SUMMARY:
120 patients age 18-64 years with dorsally displaced distal radius fractures AO-type A2, A3 and C1 are recruited from Oslo Casualty Medical Centre (Oslo Skadelegevakt). Patients are randomized to surgery with closed reduction and pins (CRPP) or open reduction and volar locking plate (VLP). The hypotheses is that CRPP will give equal function and satisfaction to VLP. Patients are followed by current practice of follow-ups until 5 weeks postoperatively, and in addition due to the study with functional tests after 2, 3, 6 and 12 months. These follow-ups will be performed by hand therapist. Scores are also recorded from Patient-Reported Wrist and Hand Evaluation (PRWHE), Quick-Dash (Q-d) and EuroQol Questionnaire (EQ-5D) questionnaires. The main efficacy measure in the study is PRWHE scores after 12 months. There will be X-ray initially, postoperatively and after 12 months. Sub-objectives in the study are analyses of cost-effectiveness (measured by EQ 5D, personnel use, use of additional healthcare service and absence from work), and differences in complications between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fractures of AO- A2, A3 and C1 which should be operated on in accordance with Norwegian guidelines
* >18 years and <65 years
* address in Oslo municipality

Exclusion Criteria:

* multitrauma
* previous fracture same wrist
* multiple injuries on the same side
* not competent to consent
* dementia / nursing home patient
* substance abuse
* foreign / tourists
* median nerve compression requiring emergency surgery
* pathological fracture
* open fracture
* congenital malformations that make it difficult to interpret data
* patient does not want surgical treatment
* not operable due to comorbidity (ASA 4, some ASA 3 after assessment by anesthesiologist)
* more than 10 days after injury

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient-Related Wrist and Hand Evaluation (PRWHE) score | 1 year
  PROM of 15 questions, score ranging from 0 (best) to 100 (worst)

SECONDARY OUTCOMES:
Quick Dash score | 1 year
  PROM of 11 questions, score ranging from 0 (best) to 100 (worst)
X-ray wrist posterior-anterior and lateral view | 1 year
  Volar tilt (degrees), radial inclination (degrees), ulnar variance (mm), stepp-off (mm)
Range of motion | 1 year
  Flexion, extension, supination and pronation measured in degrees from neutral position, pulpa palm distance in cm
Grip strength | 1 year
  Grip strength with a hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: John Williksen, MD, Study Director — Oslo University Hospital
Locations (1):
- Skadelegevakten, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No